CLINICAL TRIAL: NCT05919355
Title: BoVEL: Bo Lenger Hjemme Med Sosial Velferdsteknologi [Live Longer at Home With Social Welfare-Technology]
Brief Title: Effectiveness of a Communication Device in Home Care Services in Norway: Does Komp Make Older Adults Feel Happier, Safer and More Connected, and Able to Live Longer at Home.
Acronym: BoVEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Oslo Municipality (Other Government); No Isolation limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202916; 331810 (Other Grant/Funding Number: Research council of Norway)
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-11

CONDITIONS: Social Isolation; Well-being; Quality of Life; Mental Health; Dementia; Older Adults; Loneliness; Safety; Feeling Anxious; Technology; Home Care
Keywords: Social isolation; Komp; Communication technology; Oslo; Older adults; Home care services; Ageing in place; Gerontechnology
MeSH Terms: conditions — Social Isolation; Psychological Well-Being; Dementia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: "Intention-to-treat" (ITT)
Masking Description: There are no other parties.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Offered to try Komp (Experimental): The intervention group consists of eligible service recipients in the three boroughs, who are given the offer to try Komp. Upon receiving the offer, the participant may take up to 14 days to decide. Participants who accept, receive a Komp and use it freely; participants who decline receive services as usual. Responses are documented. Participants who accepted the offer may at any point decide to stop and return the Komp to the municipality. The actual uses and effects of the technology, being a communication technology, depends on the actions of the app users (family and friends) and platform users (care services). The investigators record the types of use and the frequency of use, but not the actual content that is transferred (e.g., pictures are counted but not seen). The investigators can also distinguish between transfers originating from the app and the platform respectively, meaning that they can analyse the effects of private and professional use separately.
  Interventions: Other: Offer to try Komp
- Services as usual (No Intervention): At a certain point, because the burrough runs out of Komp units to distribute or because they get halfway through the list, recruitment stops and no one else is offered to try Komp. All names on the burrough's list below this juncture are in the "services as normal" arm, which is the control group in this "intention-to-treat" trial. "Services as normal" means that the trial has no bearing on the participant (apart from having been informed about the project and being given the chance to opt out). They continue to receive needs-based services from their municipality, like they would have if there was no trial.

INTERVENTIONS:
Other: Offer to try Komp — The participants are offered services using the communication solution Komp. If they accept, they will receive one unit at home.
  Arms: Offered to try Komp

SUMMARY:
This study is a field trial where "Komp" is implemented and tested as part of Oslo Municipality's home care services for older adults. Komp is a "one button" communication device designed specifically for older adults who are unfamiliar with or struggle to use conventional digital technologies such as smart phones, computers, or tablets. The aim of the trial is to study the effects of increased social contact with family and care services via Komp. In a randomized design, 300 Komp units will be offered to a sample of older municipal home care service recipients. By comparing the intervention group (who are offered to test Komp for free) with the control group (who receive services as usual), the study will uncover if, on average, users of Komp 1) can live longer at home than non-users, 2) have lesser need of home care services, and 3) are happier, safer, and more socially connected.

DETAILED DESCRIPTION:
This randomized "intention-to-treat" study is a field trial where "Komp" is implemented and tested as part of Oslo Municipality's home care services for older adults.

Komp is a simple communication solution that was created by the Norwegian start-up No Isolation (ltd.) to prevent social isolation among older adults. It was designed specifically for users who are unfamiliar with or struggle to use conventional digital technologies such as smart phones, computers, or tablets. The solution consists of a screen, an app and a web-platform. The screen is a "one button" computer with a large (non-touch) screen, that can be turned on and off. As long as its on, the user can see text- or image content that have been sent to the screen from connected users, and can also receive video calls. Friends and family can connect with the screen and send pictures or messages, and make video calls, using the Komp app. Likewise, the care services can send content or make video calls using the web-based Komp platform.

The aim of the trial is to study the effects of increased social contact with family and care services via social technologies such as Komp. Specifically, the study will uncover if, on average, users of Komp 1) can live longer at home than non-users, 2) have lesser need of home care services, and 3) are happier, safer, and more socially connected. In doing so, the project will contribute systematic knowledge to facilitate evidence-based initiatives focused on social needs of older adults and the public health benefits of human interaction.

In a randomized design, 300 Komp units will be offered to a sample of older municipal home care service recipients in three Oslo boroughs. Based on the eligibility criteria (67+, recipient of municipal home care services), a recruitment list was compiled in each borough and randomized. The procedure was as follows: A search-algorithm was created to identify eligible participants. Jointly and under supervision, the boroughs applied the search-algorithm and compiled lists of service recipients. The resulting lists were then randomized under supervision. Because the three boroughs had uneven numbers of eligible inhabitants - boroughs A and B had more than twice the number of the smallest, C (N=234) - the procedure yielded disproportionately sized lists. To ensure equal chance in being offered a Komp across boroughs, the list size and number of Komp units were adjusted. C was given 60 Komp units to distribute among a randomized list of 234 eligible inhabitants, whereas boroughs A and B were each given 120 units to distribute among a randomized list of 468 of their eligible inhabitants.

Local project coordinators in each burrough systematically recruited participants by offering Komp to all names on the randomized list, working down from the top. The investigators register responses. In some instances no offer can be given, either because the participants have died or because they have moved to a care facility in the burrough or away from the burrough. In these cases, the investigators register this and move on to the next name. To avoid bias, however, these participants are included in the intervention group (as the control group will also contain participants who have died or moved during the study).

When all Komp units are distributed, or when a burrough has offered Komp to half its list, recruitment stops. All names up until then are in the intervention group; all remaining names on the list are in the control group. By comparing the intervention group (who are offered to test Komp for free) from the control group (who receive services as usual), the study will investigate if, on average, users of Komp 1) can live longer at home than non-users, 2) have lesser need of home care services, and 3) are happier, safer, and more socially connected.

ELIGIBILITY:
Inclusion Criteria:

* Must be a recipient of municipal home care services
* Must dwell in a private home (i.e., not in a permanent care or nursing home)
* Must have a registered address in one of the three burroughs

Exclusion Criteria:

- Must not score 1 on all of the following "IPLOS variables", as assessed by the municipal services: "mobility outdoors", "memory", and "cooking". IPLOS stands for Individual-based nurse and care statistics ["Individbasert pleie- og omsorgsstatistikk"], and the IPLOS variables are a set of officially sanctioned variables, the assessment of which are supposed to help municipal health and care services ascertain whether a person's performance of various functions suggests the need of assistance. Level 1 is the lowest level, meaning that there are no problems concerning this function. In a pre-study of historical data from one of the municipalities, scoring 1 on all these three variables correlated strongly with a low risk of moving to a long term care facility. By excluding them, the investigators increase the relative number of decisions to move to a long-term care facility within the study period.

Min Age: 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1114 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of days participants live at home | From the date participants were given a decision to receive home care services to the date when the participant dies, moves to a care facility, or up to a maximum of 24 months.
  The main outcome concerns the number of days elapsed from the day each participant first received municipal care services, to the day they die or move to a care facility, or when the study ends.

SECONDARY OUTCOMES:
Amount and type of care services received | From enrollment and up to 24 months.
  A secondary outcome measure concerns the level and type of care services the participants need. The investigators will record both the amount of time and the types of service that individual participants receive and how it correlates with Komp use.

OTHER OUTCOMES:
Participants' feelings of safety | Assessment happens at one point between enrollment and up to 18 months after.
  Participants are asked to self-assess their feelings of safety using a standardized scale.
Participants' social connectedness | Assessment happens at one point between enrollment and up to 18 months after.
  Participants' level and satisfaction with their social contentedness are measured using a standardized scale. In addition, the activity on the Komp is measured for Komp users.
Participants' feelings of loneliness | Assessment happens at one point between enrollment and up to 18 months after.
  Participants are asked to self-assess their feelings of loneliness using a standardized scale.
Participants' self-assessed quality of life | Assessment happens at one point between enrollment and up to 18 months after.
  Participants are asked to self-assess their overall quality of life using a standardized scale.
Participants' difficulties remembering | Assessment is supposed to happen routinely every three months, from enrollment and up to 18 months after.
  Care service providers are routinely asked to assess how much service recipients struggle to remember everyday things, on a scale of 1-5. The investigators will compare measures over time.
Participants' difficulties taking care of their health | Assessment is supposed to happen routinely every three months, from enrollment and up to 18 months after.
  Care service providers are routinely asked to assess how much service recipients struggle to take care of their health, on a scale of 1-5. The investigators will compare measures over time.

CONTACTS AND LOCATIONS:
Locations (3):
- Norway (3):
  - Oslo Municipality, Borough 4 St. Hanshaugen, Oslo
  - Oslo Municipality, Borough 13 Østensjø, Oslo
  - Oslo Municipality, Borough 14 Nordstrand, Oslo

IPD SHARING:
Plan to Share IPD: No